CLINICAL TRIAL: NCT02980367
Title: Comparison of the Clinical and Cost Effectiveness of Two Management Strategies for Non-acute Anterior Cruciate Ligament (ACL) Injury: Rehabilitation Versus Surgical Reconstruction.
Brief Title: ACL SNNAP Trial: ACL Surgery Necessity in Non Acute Patients
Acronym: ACL SNNAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12096
Record Dates: First submitted 2016-11-17; First posted 2016-12-02 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2020-11

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Anterior Cruciate Ligament; ACL; Anterior Cruciate Ligament deficiency; ACL deficiency; ACLD; Anterior Cruciate Ligament reconstruction; ACL reconstruction; Anterior Cruciate Ligament physiotherapy; Anterior Cruciate Ligament rehabilitation; ACL physiotherapy; ACL rehabilitation; Anterior Cruciate Ligament management; ACL management
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Rehabilitation; Physical Therapy Modalities; Conservative Treatment; Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACL Rehabilitation Group (Experimental): Non-surgical management [Rehabilitation] with option for later Anterior Cruciate Ligament (ACL) reconstruction, only if required.
  Interventions: Other: Non-Surgical Management (Rehabilitation)
- ACL Reconstruction Group (Active Comparator): Surgical Management - Anterior Cruciate Ligament (ACL) reconstruction surgery
  Interventions: Procedure: Surgical Management (Reconstruction)

INTERVENTIONS:
Other: Non-Surgical Management (Rehabilitation) — Routine ACL rehabilitation protocols used at the participating site will be followed. As part of the site selection process, documentary evidence of the use of or willingness to adopt a rehabilitation protocol that reflects the guidelines of the mandatory aims/goals set for the study rehabilitation intervention will be required.
  Other Names: Physical Therapy; Physiotherapy; Conservative Rehabilitation; Conservative Management
  Arms: ACL Rehabilitation Group
Procedure: Surgical Management (Reconstruction) — All surgical reconstructions will be patella tendon or hamstrings tendon depending on the surgeon's preference. All other care will be routine, including immediate post-operative care.
  Other Names: ACL Reconstruction; ACLR; ACL surgery; Anterior Cruciate Ligament Surgery; Surgical Management
  Arms: ACL Reconstruction Group

SUMMARY:
The primary objective of this study is to determine in patients with non-acute Anterior Cruciate Ligament Deficiency (ACLD) whether a strategy of non-surgical management [Rehabilitation] (with option for later ACL reconstruction, only if required) is more clinically effective and cost effective than a strategy of surgical management [Reconstruction].

DETAILED DESCRIPTION:
The ACL SNNAP study is a pragmatic multi-centre randomised controlled trial with two-arm parallel groups and 1:1 allocation ratio to compare non-surgical management (Rehabilitation) and surgical management (Reconstruction) options for patients with a symptomatic non-acute ACL deficient knee.

The objective is to determine, in patients with non-acute Anterior Cruciate Ligament Deficiency (ACLD), whether non-surgical treatment (with the option for later ACL reconstruction if required) is more effective than surgical ACL reconstruction (as measured by the Knee Injury and Osteoarthritis Outcome Score [KOOS4] at 18 months from randomisation).

Target sample size is 320 patients recruited from approx. 30 NHS orthopaedic units.

An internal pilot will be conducted with clear progression criteria regarding recruitment.

Both interventions are routine NHS treatments. Intervention content is based on a minimal set of pre-established criteria in order to ensure the integrity of the comparison while allowing for varying in practice in delivering the interventions between both surgeons and physiotherapists. This largely pragmatic approach will allow clinical management to reflect current practice and resource use within the NHS thus aiding generalisation.

Other than the allocated intervention, both groups will be followed-up in the same way to exclude bias. Follow up for study purposes will be by patient self-reported questionnaire completed using an electronic data capture collection system (a postal option will also be available). The questionnaire will include the outcomes indicated in section 4 and will be completed by participants at baseline, 6, 12 and 18 months. Non-response will be minimised through use of multiple reminders such as web based, phone and text.

Neither participants nor health care practitioners (surgeons and physiotherapists) can be blinded to receipt of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Symptomatic ACL deficiency of the native ligament1 (instability-episodes of frank giving way or feeling unstable) with ACL deficiency (either partial or complete tear) confirmed using clinical assessment and MRI scan.

Exclusion Criteria:

* Acute phase of primary ACL injury i.e. not recovered from any acute symptoms relating to their initial ACL injury.
* Previous knee surgery (other than diagnostic arthroscopy or partial meniscectomy) to index knee concomitant severe injury to contra-lateral knee.
* Meniscal pathology with characteristics that indicate immediate surgery i.e. locked knee, large bucket handle or complex cartilage tear producing mechanical symptoms.
* Knee joint status of grade 3 or 4 on the Kellgren and Lawrence scale,
* Grade 3 MCL/LCL injury, associated PCL/PLC injury
* Inflammatory arthropathy.
* Pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS4) | 18 months post randomisation
  The score is derived from 4 of 5 subscales; pain, symptoms, difficulty in sports and recreational activities, knee related quality of life.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At baseline and at 6, 12 and 18 months post randomisation
  All 5 subscales of the KOOS will be included (the fifth scale being activities of daily living).
  Anterior Cruciate Ligament Quality of Life Score (ACL-QOL)
Modified Tegner scale | At baseline and at 6, 12 and 18 months post randomisation
  Activity level will be assessed using the Modified Tegner scale, graded from 1 (low activity levels) to 10 (professional level).
Intervention related complications | At 6, 12 and 18 months post randomisation
  Any complications associated with undergoing ACL deficiency treatment will be recorded. This includes; for surgery group; re-admission, delayed hospital discharge, infection, unexpected poor range of movement (stiffness), excess bleeding, continued swelling, episodes of giving way, continued feeling of instability. For non-surgical group; continued swelling, episodes of giving way.
EuroQol EQ-5D-5L | At baseline and at 6, 12 and 18 months post randomisation
  Generic quality of life (self-reported outcome measure covering 5 health domains and used to facilitate the calculation of Quality Adjusted Life Years in health economic evaluations).
Resource-usage data | 18 months post randomisation
  Detailed resource use data on initial treatments received (surgical reconstruction or rehabilitation) and on subsequent healthcare contacts including re-operations (surgery arm), subsequent surgical reconstructions (rehabilitation arm), surgery-related complications, further rehabilitation, and primary care and other secondary care contacts out to 18 months post-randomisation. In addition, data will be collected on ability to work (e.g. sickness absences/return to work number of days off work and subjective working ability).
Anterior Cruciate Ligament Quality of Life score (ACL-QOL) | At baseline and at 6, 12 and 18 months post randomisation
  Expectations of return to activity and confidence in relation to the knee.
Patient satisfaction | At baseline and at 6, 12 and 18 months post randomisation
  Simple Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: David Beard, DPhil, Principal Investigator — University of Oxford
Locations (32):
- United Kingdom (32):
  - Betsi Cadwaladr University Health Board, Bangor
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon
  - North Bristol NHS Trust, Bristol
  - Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - Countess of Chester Hospital NHS Foundation Trust, Chester
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Frimley Health NHS Foundation Trust, Frimley
  - Royal Surrey County Hospitals NHS Foundation Trust, Guildford
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester, Leicester
  - Kings College Hospital NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Royal Berkshire NHS Foundation Trust, Reading
  - Salisbury NHS Foundation Trust, Salisbury
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Frimley Health NHS Foundation Trust, Slough
  - Stockport NHS Foundation Trust, Stockport
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Abertawe Bro Morannwg University Health Board, Swansea
  - Great Western Hospitals NHS Foundation Trust, Swindon
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - Royal Cornwall Hospitals NHS Trust, Truro
  - The Mid Yorkshire Hospitals NHS Trust, Wakefield
  - Warrington and Halton Hospitals NHS Foundation Trust, Warrington
  - Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan
  - Betsi Cadwaladr University Health Board, Wrexham
  - Yeovil District Hospital NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beard DJ, Davies L, Cook JA, Stokes J, Leal J, Fletcher H, Abram S, Chegwin K, Greshon A, Jackson W, Bottomley N, Dodd M, Bourke H, Shirkey BA, Paez A, Lamb SE, Barker KL, Phillips M, Brown M, Lythe V, Mirza B, Carr A, Monk P, Areia CM, O'Leary S, Haddad F, Wilson C, Price A; ACL SNNAP Study Group. Comparison of surgical or non-surgical management for non-acute anterior cruciate ligament injury: the ACL SNNAP RCT. Health Technol Assess. 2024 Jun;28(27):1-97. doi: 10.3310/VDKB6009. PMID 38940695
- [Derived] Beard DJ, Davies L, Cook JA, Stokes J, Leal J, Fletcher H, Abram S, Chegwin K, Greshon A, Jackson W, Bottomley N, Dodd M, Bourke H, Shirkey BA, Paez A, Lamb SE, Barker K, Phillips M, Brown M, Lythe V, Mirza B, Carr A, Monk P, Morgado Areia C, O'Leary S, Haddad F, Wilson C, Price A; ACL SNNAP Study Group. Rehabilitation versus surgical reconstruction for non-acute anterior cruciate ligament injury (ACL SNNAP): a pragmatic randomised controlled trial. Lancet. 2022 Aug 20;400(10352):605-615. doi: 10.1016/S0140-6736(22)01424-6. PMID 35988569
- [Derived] Davies L, Cook J, Leal J, Areia CM, Shirkey B, Jackson W, Campbell H, Fletcher H, Carr A, Barker K, Lamb SE, Monk P, O'Leary S, Haddad F, Wilson C, Price A, Beard D. Comparison of the clinical and cost effectiveness of two management strategies (rehabilitation versus surgical reconstruction) for non-acute anterior cruciate ligament (ACL) injury: study protocol for the ACL SNNAP randomised controlled trial. Trials. 2020 May 14;21(1):405. doi: 10.1186/s13063-020-04298-y. PMID 32410697